CLINICAL TRIAL: NCT04946968
Title: A Phase II Multi-Centre Study Evaluating the Efficacy of Dacomitinib for Patients With Epidermal Growth Factor Receptor (EGFR)-Driven Advanced Solid Tumours With Low EGFR-AS1 IncRNA Expression or Other Novel Emerging Biomarkers
Brief Title: Phase-2 Dacomitinib Study on Patients With EGFR-Driven Advanced Solid Tumours With Low EGFR-AS1 IncRNA Expr or Other Novel Emerging Biomarkers
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Centre, Singapore (Other)
Collaborators: Singapore Translational Cancer Consortium (Unknown); Cancer Science Institute of Singapore (Unknown); Genome Institute of Singapore (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STCC-01
Record Dates: First submitted 2021-06-21; First posted 2021-07-01 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Advanced Solid Tumours; Non-small Cell Lung Cancer; Head and Neck Squamous Cell Carcinoma
Keywords: EGFR-driven advanced solid tumours; Low EGFR-AS1 lncRNA expression; Novel emerging biomarker
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Squamous Cell Carcinoma of Head and Neck | interventions — dacomitinib

STUDY DESIGN:
Intervention Model Description: Eligible subjects will be allocated to one of four cohorts based on tumour type and presence of specific biomarker. All subjects in cohorts 1 to 3 will have tumours that demonstrate low EGFR-AS1 lncRNA expression as determined through a companion diagnostic biomarker suite (consisting of three components - EGFR Q787Q AA genotype, low AS1 lncRNA levels and increased EGFR isoform D/A ratio).
  * Cohort 1 will consist of squamous NSCLC patients with the presence of at least 1 out of 3 in the biomarker suite.
  * Cohort 2 will consist of HNSCC patients with the presence of at least 1 out of 3 in the biomarker suite.
  * Cohort 3 will consist of any other solid tumour with the presence of at least 1 out of 3 in the biomarker suite.
  * Cohort 4 will have tumours that demonstrate the presence of a novel emerging biomarker including but not limited to NRG1 fusions and specific MET SNPs.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dacomitinib (Experimental): Oral Dacomitinib tablets, once daily.
  Interventions: Drug: Oral Dacomitinib

INTERVENTIONS:
Drug: Oral Dacomitinib — All subjects will receive the open-label Dacomitinib as tablets for oral self-administration on a continuous daily basis at a dose of 30 mg for one cycle. For subjects eligible for dose titration after Cycle 1, and after shared patient and investigator decision, these subjects will receive Dacomitinib 45 mg orally on a continuous daily basis.

SUMMARY:
Eligible subjects will be allocated to one of four cohorts based on tumour type and presence of specific biomarker.

Subjects will receive open-label Dacomitinib as tablets for oral administration on a continuous daily basis at a dose of 30 mg for one cycle. After one cycle, a toxicity assessment will be conducted. Subjects with >=G2 toxicity attributable to dacomitinib, will continue dacomitinib at 30 mg orally once daily.

In subjects with <=G1 toxicity, investigator and subjects will make a shared decision for dose escalation of dacomitinib to 45 mg orally once daily or continuation of dacomitinib at 30 mg orally once daily. Subjects will then continue on therapy until disease progression, new systemic anticancer therapy instituted, intolerable toxicities, withdrawal of consent, death, or investigator decision dictated by protocol compliance, whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

* Provision of a voluntarily given, personally signed and dated, written informed consent document. If consent cannot be expressed in writing, it must be formally documented and witnessed, ideally via an independent trusted witness;
* Age ≥ 21 years, male or female;
* Documentation of the presence of low EGFR-AS1 lncRNA expression as determined using the specifically designed companion diagnostic biomarker suite provided by the Sponsor (cohorts 1 to 3) or the presence of a novel emerging biomarker of EGFR family pathway addiction as determined by the Sponsor (cohort 4);
* Study cohorts:

  * Cohort 1: advanced or metastatic EGFR wildtype squamous NSCLC, after progression on or after, or intolerance to, one or more lines of standard of care (SOC) therapy, per local SOC guidelines. In subjects without an activating oncogenic driver mutation, after progression on or after, or intolerance to, platinum-containing combination chemotherapy. In subjects harbouring an activating oncogenic driver mutation, after progression on one or more SOC mutation-targeting TKI, per local SOC guidelines, or for whom no SOC mutation-targeting TKI is available. TKI therapy need not be the most recent prior therapy. Subjects harbouring an activating EGFR mutation are not eligible;
  * Cohort 2: advanced or metastatic head and neck squamous cell carcinoma, after progression on or after, or intolerance to, platinum-containing combination chemotherapy. This need not be the most recent or prior regimen;
  * Cohort 3: all advanced or metastatic solid tumours (excluding squamous NSCLC and HNSCC), after progression on or intolerance to at least one line of SOC therapy per local guidelines;
  * Cohort 4: all advanced or metastatic solid tumours, after progression on or intolerance to at least one line of SOC therapy per local guidelines;
* Have an ECOG PS of ≤2;
* Life expectancy of at least 3 months;
* Site of disease amenable to biopsy and be a candidate for tumour biopsy according to the treating institution's own guidelines and requirements for such procedure. Subjects must be willing to undergo a tumour biopsy at screening, and on treatment on this study;
* Radiologically measurable disease by RECIST v1.1 criteria:

  * At least one target lesion that has not previously been radiated and is measurable according to RECIST v1.1;
  * Acceptable radiologic procedures for disease assessment include contrast enhanced conventional or spiral computed tomography (CT), or contrast enhanced magnetic resonance imaging (MRI);Non contrast CT scan is acceptable only for subjects who are both allergic to intravenous contrast and unable to cooperate with MRI, or MRI is not available. The following are not allowed as sole documentation of target lesions: CT component of a positron emission tomography (PET)/CT, ultrasound alone, nuclear scans (including bone or PET scans), chest X-ray or bone radiographs, and tumour markers;
* Adequate organ function, including:

  * Estimated creatinine clearance ≥30 mL/min (as determined by Cockcroft-Gault formula or the study site's standard formula);
  * Absolute neutrophil count (ANC) ≥1500 cells/mm3;
  * Platelets ≥100,000 cells/mm3;
  * Hemoglobin ≥10.0 g/dL;
  * Bilirubin ≤1.5 x upper limit of normal (ULN);
  * Aspartate aminotransferase (AST; also known as SGOT) and Alanine aminotransferase (ALT; also known as SGPT) ≤2.5 x ULN (≤5.0 x ULN if hepatic metastases).
* Female subjects must be postmenopausal (defined as 12 months of amenorrhea following last menses), or they or their partners must be surgically sterile, or must agree to use effective contraception while receiving study treatment and for at least 3 months thereafter. The definition of effective contraception will be based on the judgment of the investigator using following criteria:

  * Acceptable contraception for women include implants, injectables, combined oral contraceptives, intrauterine devices (IUDs), sexual abstinence, or a partner who has been surgically sterile (e.g. by vasectomy) for at least 6 months. Acceptable contraception for a male includes surgical sterility (e.g. by vasectomy) for at least 6 months, sexual abstinence, or condoms plus spermicide.
* All female subjects with reproductive potential must have a negative pregnancy test (serum or urine) before starting study treatment;
* Male subjects or their female partners must be surgically sterile or must agree to use effective contraception while receiving study treatment and for at least 3 months thereafter. The definition of effective contraception will be based on the judgment of the investigator. Or female partners must be postmenopausal (defined as 12 months of amenorrhea following last menses);
* Willing and able to comply with study scheduled visits, treatment plans, laboratory tests, and other study procedures.

Exclusion Criteria:

* Subjects with symptomatic brain metastases or leptomeningeal metastases who are neurologically unstable or require increasing doses of steroids to manage central nervous system (CNS) symptoms within two weeks prior to starting dacomitinib;
* Any surgery (not including minor procedures such as lymph node biopsy), palliative radiotherapy or pleurodesis within 2 weeks of baseline assessments;
* Any clinically significant gastrointestinal abnormalities that may impair intake, transit or absorption of the study drug, such as the inability to take oral medication;
* Current enrollment in another therapeutic clinical study;
* Any psychiatric or cognitive disorder that would limit the understanding or rendering of informed consent and/or compromise compliance with the requirements of this study or known drug abuse/alcohol abuse;
* History of, or currently suspected, diffuse non-infectious pneumonitis or interstitial lung disease including:

  * Past medical history of interstitial lung disease, drug-induced interstitial disease, radiation pneumonitis which required steroid treatment or any evidence of clinically active interstitial lung disease;
  * Pre-existing idiopathic pulmonary fibrosis evidenced by CT scan at baseline;
  * Insufficient lung function as determined by either clinical examination or an arterial oxygen tension of <70 Torr.
* Any history of galactose intolerance, Lapp lactase deficiency or glucose-galactose malabsorption;
* Clinically important abnormalities in cardiac rhythm, conduction or morphology of resting ECG (e.g. complete left bundle branch block, second degree heart block, third degree heart block) OR:

  * Diagnosed or suspected congenital long QT syndrome;
  * Any history of clinically significant ventricular arrhythmias (such as ventricular tachycardia, ventricular fibrillation, or Torsades de pointes);
  * Prolonged QTc interval on electrocardiogram (ECG); QTc must be less than CTCAEv5.0 Grade 2 (≤480 msec) using Fridericia's or Bazett's correction formula with a manual reading by the investigator if required. The ECG may be repeated for evaluation of eligibility after management of correctable causes for observed QTc prolongation;
  * Any history of second- or third-degree heart block;
  * Heart rate <45 beats per minute on ECG in the presence of clinical symptoms (e.g., hypotension, evidence of hypoperfusion);
* Severely impaired (defined as Child-Pugh Class C) hepatic dysfunction;
* Prior malignancy: Subjects will not be eligible if they have history of, or evidence of another concurrent malignancy within 2 years prior to registration. Exception would be effectively treated past history of non-melanoma skin cancer or in-situ cervical cancer with no evidence of active disease. Patients with a history of other malignancies are eligible if they have been continuously disease free for at least 2 years after definitive primary treatment;
* Other severe acute or chronic medical condition that may increase the risk associated with study participation or study drug administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the subject inappropriate for entry into this study;
* Use of narrow therapeutic index drugs that are CYP2D6 substrates (procainamide, pimozide, and thioridazine etc.) from screening to randomization.
* Active primary immunodeficiency, known HIV infection, or known active hepatitis B or C infection. Subjects with past or resolved hepatitis B virus (HBV) infection are eligible if:

  * Hepatitis B surface antigen (HBsAg) negative and hepatitis B core antibody [anti-HBc] positive; OR
  * HBsAg positive and HBV deoxyribonucleic acid (DNA) viral load is documented to be ≤2000 IU/mL in the absence of anti-viral therapy and during the previous 12 weeks prior to the viral load evaluation with normal transaminases; OR
  * HBsAg positive and HBV DNA viral load is documented to be ≤2000 IU/mL in the absence of anti-viral therapy and during the previous 12 weeks prior to the viral load evaluation with liver metastasis and abnormal transaminases alanine aminotransferase (ALT)/ aspartate aminotransferase (AST) <3 upper limit of normal (ULN)
  * Subjects with a history of hepatitis C infection will be eligible for enrolment only if the viral load according to local standards of detection is documented to be below the level of detection in the absence of anti-viral therapy during the previous 12 weeks (i.e., sustained viral response according to the local product label but no less than 12 weeks, whichever is longer) prior to the viral load evaluation.

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2021-08-24 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate | From time of first study drug administration until first occurrence of disease progression, up to 36 months.
  The proportion of subjects with a BOR of either CR or PR, where BOR is the best response recorded from the start of treatment until disease progression.

SECONDARY OUTCOMES:
Progression Free Survival | The time from start of treatment to the date of disease progression as defined by RECIST v1.1 per investigator review or death due to any cause, whichever occurs first, up to 36 months.
  The time from start of treatment to the date of disease progression or death due to any cause, whichever occurs first.
Duration of Response | The time from the initial response to therapy to the date of subsequent disease progression as defined by RECIST v1.1 per investigator review or date of death (if cause of death is due to PD), whichever earlier, up to 36 months.
  The time from the initial response to therapy to the date of subsequent disease progression or date of death (if cause of death is due to PD), whichever earlier.
Overall Survival | The time from start of treatment to the date of death for any cause, up to 36 months.
  The time from start of treatment to the date of death for any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel SW Tan, Principal Investigator — National Cancer Centre, Singapore; Boon Cher Goh, Principal Investigator — National University of Singapore
Locations (2):
- Singapore (2):
  - National University Cancer Institute, Singapore, Singapore
  - National Cancer Centre Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No